CLINICAL TRIAL: NCT01286974
Title: Disposition of [14C]ABT-869 in Patients With Solid Tumors Following a Single Oral Dose Administration
Brief Title: A Pharmacokinetic Study to Access How the Body Absorbs and Removes Linifanib in Male Patients With Advanced Solid Tumors.
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated early, Sponsor Decision
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: M10-966
Record Dates: First submitted 2011-01-28; First posted 2011-02-01 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — linifanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ADME (Experimental): [14C]linifanib
  Interventions: Drug: [14C]linifanib
- Extension (Experimental): linifanib
  Interventions: Drug: ABT-869, linifanib

INTERVENTIONS:
Drug: [14C]linifanib — [14C]linifanib, single administration, oral liquid
  Arms: ADME
Drug: ABT-869, linifanib — linifanib once a day (QD), oral tablet
  Arms: Extension

SUMMARY:
A pharmacokinetic study to access how the body absorbs and removes linifanib in male patients with advanced solid tumors.

DETAILED DESCRIPTION:
This study is designed to assess the mass balance of [14C]linifanib and the metabolic profiles of linifanib in 4 subjects with advanced solid tumors following a single oral dose. Subjects may continue on linifanib after completion of the metabolism study. The results of this study will determine the exposure of major metabolites and excretion pathway(s) of the parent drug and metabolites of linifanib in humans.

ELIGIBILITY:
Inclusion Criteria

* Subject must be >/= 18 years of age.
* Subject must have a histologically or cytologically confirmed non-hematologic malignancy.
* Eastern cooperative Oncology Group (ECOG) Performance Score of 0 to 2.
* Subject must have adequate bone marrow, renal and hepatic function.
* Subject must have Partial Thromboplastin Time (PTT) </= 1.5 x Upper Limit of Normal (ULN) and International Normalized Ratio (INR) </= 1.5.
* Subject must be capable of understanding and complying with parameters as outlined in the protocol and able to sign the informed consent.

Exclusion Criteria

* Subject has received previous administration of a radiolabeled research substance within 12 months prior to Study Day 1 or exposure to significant radiation (e.g., barium meal, etc.) within the past 3 months or within a period defined by 5 half-lives, whichever is shorter, prior to Study Day 1.
* Subject has received anti-cancer therapy including investigational agents, cytotoxic chemotherapy, radiation, hormonal or biologic therapy within 21 days or within a period defined by 5 half-lives, whichever is shorter, prior to Study Day 1.
* Subject is currently using a known inhibitor (e.g., ketoconazole) or inducer (e.g., rifampin) of cytochrome P450 3A (CYP3A) within 1 month prior to Study Day 1.
* Subject has not recovered to less than or equal to grade 1 clinically significant adverse effects/toxicities of the previous therapy.
* Subject has undergone major surgery within 21 days of Study Day 1.
* The subject has brain or meningeal metastases.
* The subject has non-small cell lung cancer (NSCLC) with a predominant squamous cell histology.
* Subject is receiving therapeutic anticoagulation therapy.
* Subject has a history of/or currently exhibits clinically significant events of bleeding (e.g., hemoptysis).
* Subject has proteinuria Common Terminology Criteria (CTC) Grade > 2 at baseline.
* Subject currently exhibits symptomatic or persistent, uncontrolled hypertension.
* Subject has a history of myocardial infarction within 6 months.
* Subject has known autoimmune disease with renal involvement.
* Subject is receiving combination anti-retroviral therapy for human immunodeficiency virus (HIV).
* Clinically significant uncontrolled conditions/medical symptoms.
* Subject has a documented left ventricular (LV) ejection fraction < 50%.
* Subject has previously received linifanib.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic Profile | Various timepoints from Day 1 through approximately Day 9
  Blood samples for the pharmacokinetics (PK) of linifanib will be collected at designated time points.
Total radioactivity | Various timepoints from Day 1 through approximately Day 9
  Blood, urine, and fecal samples for total radioactivity analysis will be collected at designated time points.

SECONDARY OUTCOMES:
Safety (Number of subjects with adverse events and/or dose-limiting toxicities) | At each treatment visit (daily for first 9 days and then approximately every 4 weeks through end of treatment)
  Adverse event monitoring, lab test assessments, physical exam and vital signs will be evaluated throughout the study.

CONTACTS AND LOCATIONS:
Overall Officials: Mark D. McKee, MD, Study Director — Abbott
Locations (2):
- United States (2):
  - Site Reference ID/Investigator# 40942, Cleveland, Ohio
  - Site Reference ID/Investigator# 53663, Cleveland, Ohio